CLINICAL TRIAL: NCT03303170
Title: A Prospective, Multicenter, Randomized, Controlled, Evaluator-Blinded Study of the Safety and Effectiveness of Sebacia Microparticles as an Accessory to 1064 nm Nd:Yag Laser in the Treatment of Facial Inflammatory Acne Vulgaris
Brief Title: Non-Significant Risk Study of Sebacia Microparticles in the Treatment of Facial Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sebacia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEB-0493
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sebacia Microparticles (Experimental)
  Interventions: Device: Sebacia Microparticles
- Nd:Yag Laser (Active Comparator)
  Interventions: Device: Nd:Yag Laser

INTERVENTIONS:
Device: Sebacia Microparticles — Topical microparticle suspension
  Arms: Sebacia Microparticles
Device: Nd:Yag Laser — Laser delivering 1064 nm wavelength light
  Arms: Nd:Yag Laser

SUMMARY:
Prospective, randomized, controlled, parallel group clinical study with blinded assessment evaluating Sebacia Microparticles (SM) with Nd:Yag laser in facial inflammatory acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate acne vulgaris
* At least 15 inflammatory acne lesions
* Skin phototype I - III
* Able to understand and comply with study requirements

Exclusion Criteria:

* Severe acne vulgaris
* Nodulocystic acne
* Ongoing use of medications and/or treatments for acne
* New hormone regimen (used for less than 12 weeks)
* Significant medical or mental health condition

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Change in number of inflammatory acne lesions | Week 12

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Clear Dermatology & Aesthetics Center, Scottsdale, Arizona
  - Scripps Health, San Diego, California
  - Miami Dermatology & Laser Institute, Miami, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Dermatology, Laser & Vein Institute, Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - International Clinical Research, Murfreesboro, Tennessee
  - Austin Institute for Clinical Research, Austin, Texas
  - The Center for Skin Research, Katy, Texas
  - Premier Clinical Research, Spokane, Washington

REFERENCES:
- See also: Sponsor Website — http://www.sebacia.com